CLINICAL TRIAL: NCT00213005
Title: A Phase 1 Safety and Acceptability Study of Carraguard® Among HIV Positive Women and Men in Durban, South Africa
Brief Title: Safety and Acceptability of Carraguard® in HIV Positive Women and Men
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Medical Research Council (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: Population Council #297
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: HIV Infections
Keywords: Microbicides; HIV prevention; HIV positive; carrageenan; safety trial; Treatment Experienced; HIV
MeSH Terms: conditions — HIV Infections; HIV Seropositivity

INTERVENTIONS:
Drug: Carraguard (PC-515)

SUMMARY:
The study objectives were to assess the mucosal safety of Carraguard® gel when applied vaginally once per day for 14 days by sexually abstinent and sexually active, HIV-positive women; to evaluate the effect of Carraguard® gel on the vaginal flora in these women; to evaluate the effect of Carraguard® gel on shedding of HIV-1 in the genital tract of these women; to evaluate the safety of Carraguard® gel when applied directly to the penis once per day for 7 days by sexually abstinent, HIV-positive men; to assess whether symptoms reported by female and male participants during the study may be related to the use of Carraguard® gel; and to examine dimensions of the acceptability of, and compliance with, the study and placebo products.

DETAILED DESCRIPTION:
We proposed a safety study of the Council's lead candidate microbicide, Carraguard® in three cohorts in Durban, South Africa: sexually abstinent HIV-positive women, sexually abstinent HIV-positive men, and sexually active HIV-positive women. Sexually active women must be in an HIV-positive seroconcordant relationship (confirmed by HIV testing of the woman and her male partner) and written informed consent was obtained from the male partners. Women and men in each cohort were randomized to one of three study groups: Carraguard® gel, its matching placebo methyl-cellulose gel, or no product.

The main objectives of this study were to investigate changes in the vulvar, vaginal, and cervical epithelia, the vaginal flora, and HIV-1 shedding in the genital tract of female participants, and changes of the penile skin and epithelia of male participants. We also evaluated symptoms reported by participants, and several dimensions of the acceptability of and compliance with the study or placebo gel. Reactions to a non-contraceptive microbicide were assessed, as well as reasons for voluntary discontinuation and non-use of Carraguard® or the placebo (determined by review of daily diary) was recorded. Exit focus group discussions were held with male and female participants to discuss aspects of acceptability and compliance. Self-reported symptoms were also investigated by clinical examination as needed and study endpoints included genital itching or burning, frequent urination, burning while urinating, genital pain, pain during sex, and abnormal vaginal or penile discharge.

ELIGIBILITY:
Inclusion Criteria:

* Positive for HIV-1 by licensed HIV test (with confirmation) and agree to be informed of the test result
* Age 18 to 45 years old, for women (no maximum age for men)
* In good health, defined as CD4+ cell count >200 x 106/L and current absence of opportunistic infections that may interfere with protocol adherence
* If on treatment for HIV infection (including immune-boosters such as Moducare and vitamins): treatment should stay constant for the duration of the study
* For sexually abstinent cohort: Willing to abstain from sexual intercourse and masturbation for the duration of the study (3 weeks) and for the 48 hours before joining the study
* For sexually active cohort: Willing to have sex with only one male partner, and male partner is willing to have sex with only the participant, for the duration of the study
* Regular menstrual cycle (3-5 weeks between periods) or amenorrheic due to long-term (three months or more) DMPA use (and have had no DMPA-related side effects that could interfere with study participation in the last 6 months)
* Planning on living in Durban for the next 6 months
* Willing to refrain from using any other vaginal products for the duration of the study (3 weeks), including other spermicides, diaphragm/cervical cap, traditional drying and tightening agents, douches, tampons, and medicinal products
* Willing and able to comply with all other aspects of the study protocol, including clinical evaluations and study gel administration (if applicable)
* Willing and able to give informed consent.

Exclusion Criteria:

* Currently pregnant, menopausal or lactating, or desire to become pregnant at the time of study participation
* Current or recent participation (within past 30 days) in any other clinical trial, including trials of HIV therapeutics and trials of vaginal products (this does not include the ongoing study in the Department of Paediatrics of King Edward VIII Hospital)
* Delivery, miscarriage or abortion within the last six weeks
* Gynecological surgery or instrumentation in the last three months
* History of non-menstrual vaginal bleeding with intercourse in the last month
* Presence of a clinically detectable genital abnormality (i.e. vulvar, vaginal, cervical and/or perianal ulcer and/or lesion) on which the epithelium is currently disrupted or is likely to disrupt (e.g. herpes blister). Women with healed/dried-up lesions from a past infection, or with a lesion on which the epithelium is currently intact or unlikely to disrupt, will be eligible for enrollment.
* Presence of a sexually transmitted infection (STI), symptomatic yeast infection, or bacterial vaginosis (BV), as diagnosed by clinical exam or laboratory testing at screening. Women with asymptomatic yeast infection or BV may be enrolled.
* Abnormal Pap smear (CIN I or higher) at screening
* Use of any spermicide or spermicidally lubricated condom within the week prior to enrollment.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60
Dates: Start 2002-06 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Safety: genital findings, epithelial disruption, vaginal flora changes, genital shedding, inflammation & self-reported symptoms. Assessments were made weekly at days 7, 14 & 21.
Acceptability: interviewer-administered questionnaires & daily diaries. Interviewer-administered questionnaires assessed at day 21 & daily diaries were assessed at days 14 and 21.

CONTACTS AND LOCATIONS:
Overall Officials: Janneke van de Wijgert, Ph.D., Principal Investigator — International Antiviral Therapy Evaluation Center; Gita Ramjee, Ph.D, Principal Investigator — Medical Research Council
Locations (1):
- Medical Research Council, Durban, South Africa

REFERENCES:
- [Derived] van de Wijgert JH, Braunstein SL, Morar NS, Jones HE, Madurai L, Strickfaden TT, Moodley M, Aboobaker J, Ndlovu G, Ferguson TM, Friedland BA, Hart CE, Ramjee G. Carraguard Vaginal Gel Safety in HIV-Positive Women and Men in South Africa. J Acquir Immune Defic Syndr. 2007 Dec 15;46(5):538-46. doi: 10.1097/qai.0b013e318159d5a8. PMID 18193495